CLINICAL TRIAL: NCT04263948
Title: Multidom Remote Monitoring of Patient With Advanced Pancreatic Cancer Treated With Florinox Using the PiCaDo Domomedecine Plateform
Brief Title: Multidom Remote Monitoring of Patient With Advanced Pancreatic Cancer Treated With Florinox Using the PiCaDo Plateform
Acronym: MULTIDOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Faculty of Medicine Paris Saclay University (Unknown); Altran (Unknown); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-12-033
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Pancreas Cancer
Keywords: pancreas cancer; Plateform monitoring; metastatic or "borderline"; telemedicine; tele monitoring; telecare; emergency hospitalisations; patient-centered medicine; internet platform; circadian rhythms; chronotherapy; physical activity; sleep; patient -reported outcomes; symptoms; quality of life; compliance; sensors; electronic questionnaires
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Motor Activity; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Picado Arm (Experimental): All the patients undergo multidimensional tele monitoring for 7 weeks using an upgraded version of the Picado internet platform
  Interventions: Device: Picado system internet platform and connected objects

INTERVENTIONS:
Device: Picado system internet platform and connected objects — The system will monitor the circadian rhythms, physical activity, sleep, symptoms and body weight of patients with advanced pancreatic cancer during one week before (baseline) and six weeks after the 1st course of standard mFOLFIRINOX. The reach of preset thresholds for several parameters that are automatically computed will trigger alerts toward approved health professionals, and their responses will be traced.

SUMMARY:
Pancreatic cancer is a rapidly developing cancer with a poor prognosis. The mFOLFIRINOX protocol has become the standard medical treatment for this pathology. However, mFOLFIRINOX is the cause of severe toxicities including leukoneutropenia, thrombocytopenia, diarrhea, nausea-vomiting, anorexia, asthenia, weight loss and peripheral sensory neuropathy. Therefore, its indication is limited to patients in good general condition. In practice, it is often interrupted upon the occurrence of hematological and/or clinical grade 3-4 toxicities, Remote patient tele-monitoring of symptoms (Patient Reported Outcomes), body weight, circadian rhythms, sleep and activity would allow the identification of early warning signals reflecting deterioration or improvement in the health of these fragile patients, and trigger proactive interventions, while they are outside the hospital. Thus, the MultiDom study proposes a comprehensive tele-monitoring and telecare strategy that would complement standard of care over a 7-weeks period to 42 consenting patients. The patients receive neoadjuvant or first line chemotherapy with mFOLFIRINOX for advanced or metastatic pancreatic cancer at one of four centres in Ile-de-France region (France).

DETAILED DESCRIPTION:
MultiDom stands up among the very first prospective patient-entered and multidimensional, multiactor and multicenter study, that assesses the qualitative and quantitative impact of mFOLFIRINOX on the daily life of patients with pancreatic cancer in real time. Main endpoint is the rate of patients undergoing toxicity-related emergency hospitalisations, and the objective is to reduce it to <10%. Telemonitored data-based proactive interventions will expectedly prevent worsening of patients 'health, and maintain their chances of disease control on effective mFOLFIRINOX chemotherapy.

Participating patients have usual follow up and treatments for their disease, but also: wear a chest sensor that measures and teletransmits accelerometry, surface temperature and 3D-orientation every min, weigh themselves daily on a BLE-balance, with immediate weight tele transmission, and fill out electronic PRO questionnaires daily using a telecommunicating tablet.

All data are tele transmitted to an approved health data hub, and automatically analysed for physical activity, sleep, circadian rhythms, symptoms scores trends in real time. Visualization screens and alerts are generated according to preset thresholds, and medical team responses are traced.

Currently recruiting centres:

1. Clinique du Mousseau, Evry, France
2. Hospital Paul Brousse (Assistance Publique-Hôpitaux de Paris), Villejuif, France
3. Clinique St-Jean L'Ermitage, Melun, France
4. Private Hospital of Antony, Antony, France

ELIGIBILITY:
Inclusion Criteria:

-Histological or cytological diagnosis of pancreatic adenocarcinoma

* Locally advanced or metastatic pancreatic cancer
* With or without previous surgery (pancreas and / or metastases)
* Performance status of 0 or 1 according to WHO
* Age between 18 and 85 years old included
* No history of prior chemotherapy or radiotherapy
* Absence of cutaneous or mucosal jaundice or skin pruritus
* No proven thrombosis
* Absence of heart disease or other pathology poorly controlled by current treatments
* Bilirubinemia and alkaline phosphatases <1.5 ULN (with or without stent)
* Hematological, renal and hepatic laboratory tests authorizing the administration of mFOLFIRINOX
* Affiliated subject or beneficiary of a social security scheme
* Patient who freely signed informed consent

Exclusion Criteria:

* Immediately resectable pancreatic cancer
* No histological or cytological evidence of pancreatic adenocarcinoma
* Performance status> 1 (WHO)
* Age <18 and> 85 years old
* Prior administration of chemotherapy or radiotherapy
* Skin jaundice and / or pruritus
* Uncontrolled venous or arterial thrombosis
* Co morbidity not controlled by a specific treatment
* Biological anomalies contraindicating the administration of one or more drugs which make up FOLFIRINOX
* Lack of GPRS coverage in the home
* Patient participating in another clinical study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, lactating or parturient woman
* Patient hospitalized without consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Toxicity-related emergency hospitalisation rate | First cycle of treatment of 6 weeks
  The main objective is to assess the toxicities occurring during the 6 weeks following the start of the 1st cycle of FOLFIRINOX in conventional administration in patients benefiting from the PiCADo telemonitoring system.
Rates and grades toxicity and early tumor responses | First cycle of treatment of 6 weeks
  Secondary objectives include rates and grades of toxicity and early tumor responses, as well as PiCADo platform performances and users perceptions.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Mousseau, Évry, IDF, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the original trial report manuscripts will be shared after deidentification. Supportive information will consist in the study protocol.
Supporting Information: Study Protocol
Time Frame: Data will be available for two years following article publication at jf.oudet@ecten.eu.
Access Criteria: Access will be granted to researchers who provide a methodologically sound proposal and only aim toward publicly available scientific publication, and in accordance with the French General Data Protection Regulation."

REFERENCES:
- [Background] Bouchahda M, Komarzynski S, Ulusakarya A, Attari A, Duprès A, Breda G, Fritsch A, Adam R, Lévi F (2020) Improving FOLFIRINOX safety in pancreatic cancer patients through multidimensional remote monitoring and proactive care using a domomedecine mobile platform. J Clin Oncol 38: TPS4673.
- [Background] Levi F, Komarzynski S, Huang Q, Young T, Ang Y, Fuller C, Bolborea M, Brettschneider J, Fursse J, Finkenstadt B, White DP, Innominato P. Tele-Monitoring of Cancer Patients' Rhythms during Daily Life Identifies Actionable Determinants of Circadian and Sleep Disruption. Cancers (Basel). 2020 Jul 17;12(7):1938. doi: 10.3390/cancers12071938. PMID 32708950
- [Background] Innominato P, Komarzynski S, Karaboue A, Ulusakarya A, Bouchahda M, Haydar M, Bossevot-Desmaris R, Mocquery M, Plessis V, Levi F. Home-Based e-Health Platform for Multidimensional Telemonitoring of Symptoms, Body Weight, Sleep, and Circadian Activity: Relevance for Chronomodulated Administration of Irinotecan, Fluorouracil-Leucovorin, and Oxaliplatin at Home-Results From a Pilot Study. JCO Clin Cancer Inform. 2018 Dec;2:1-15. doi: 10.1200/CCI.17.00125. PMID 30652550
- [Derived] Bouchahda M, Ulusakarya A, Thirot-Bidault A, Attari A, Bossevot R, Tuligenga R, Hammel P, Adam R, Levi F. Multicentre, interventional, single-arm study protocol of telemonitored circadian rhythms and patient-reported outcomes for improving mFOLFIRINOX safety in patients with pancreatic cancer (MultiDom, NCT04263948). BMJ Open. 2023 Jun 7;13(6):e069973. doi: 10.1136/bmjopen-2022-069973. PMID 37286324